CLINICAL TRIAL: NCT00289939
Title: Reducing HIV & Domestic Violence Risk in Women Offenders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Multnomah County Health Department (Other Government)
Collaborators: Oregon Department of Human Services (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01DA012572 (NIH)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2006-02-28 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections; Domestic Violence; Sexually Transmitted Diseases
Keywords: women; women's health; HIV; risk factors; risk behaviors; prevention; motivational interviewing; domestic violence; partner violence; behavioral trial; community justice; criminal justice
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Risk-Taking | interventions — Seroconversion

INTERVENTIONS:
Behavioral: Motivational interviewing to reduce risk for HIV and DV

SUMMARY:
The long-term goal of this work is to reduce the prevalence of HIV and domestic violence among women at risk by encouraging self-protective behaviors. To obtain this goal, Multnomah County Health Department and Oregon Department of Human Services have conducted a randomized trial of an intervention to prevent HIV and domestic violence among women who have recent criminal justice involvement and who are at risk for HIV infection.

Women enrolled in the study were randomly assigned to one of three study conditions:

* Group 1: these women received information on local resources addressing HIV prevention, domestic violence, and life stability issues; they did not receive any counseling sessions as part of the study itself.
* Group 2: these women received up to ten supportive counseling sessions based on the techniques of motivational interviewing. These sessions aimed to reduce HIV risk and to improve life stability.
* Group 3: these women received up to ten supportive counseling sessions based on motivational interviewing. These sessions aimed to reduce risk for HIV and domestic violence and to improve life stability.

The primary hypotheses of this study were:

* 1. Supportive counseling (motivational interviewing) addressing HIV prevention and increased life stability will lead to reductions of HIV risk behavior among women enrolled in the study.
* 2. Supportive counseling (motivational interviewing) addressing domestic violence prevention, HIV prevention, and increased life stability, will bring about reductions in experiences of domestic violence and a reduction of HIV risk among these women.
* 3. The supportive counseling received in this study will enhance these women's self-efficacy, self-esteem, and psychological well-being.

Women in all three experimental groups were interviewed at the beginning of the study and again after 4, 7, and 10 months. These assessment interviews asked questions about: HIV risk; experiences of domestic violence; and life stability issues such as education, employment, and housing; and included biological testing for HIV and sexually transmitted diseases. Women in Group 2 and Group 3 participated in up to 10 sessions of supportive counseling (motivational interviewing) between the time of enrollment and the 4-month interviews.

ELIGIBILITY:
Inclusion Criteria:

* women
* who were 18 years or older
* who had been in jail or prison in the past year or who were currently on parole or probation
* who had engaged in HIV-related risk behaviors (injection drug use, crack use, intercourse with a male injection drug user, exchanging sex, or having had ten or more sexual partners) in the past year

Exclusion Criteria: Women were excluded from the study if:

* they were unable to give informed consent
* they were HIV positive at the time of screening for enrollment
* they reported highly unstable living conditions at screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 530
Dates: Start 2000-09; Study Completion 2005-01

PRIMARY OUTCOMES:
unprotected sex
injection drug use
intimate partner violence
violence from others

SECONDARY OUTCOMES:
self-esteem
anxiety
depression
housing stability
employment
education

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Stark, Ph.D., Principal Investigator — Multnomah County Health Department
Locations (1):
- SE Health Center, Portland, Oregon, United States